CLINICAL TRIAL: NCT07316218
Title: Personalized Wearable Robotics for Upper-limb Motor Rehabilitation in Neurological Patients. A Pilot Study.
Acronym: RONDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico Posteraro (Other)
Collaborators: Scuola Superiore Sant'Anna di Pisa (Other)
Responsible Party: Sponsor-Investigator, Federico Posteraro, Head of Rehabilitation Department, Azienda USL Toscana Nord Ovest
Organization: Azienda USL Toscana Nord Ovest (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: RONDA201813581; PAR FAS 2007-2013 (Other Grant/Funding Number: MIUR - MISE - REGIONE TOSCANA DGRT 758/2013)
Record Dates: First submitted 2025-11-17; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Stroke
Keywords: Stroke; Pilot Study; Exoskeleton
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Traditional feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NESM-alpha (Experimental): Patients with severe or moderate upper-limb motor impairment (UEFM ≤ 42) receive 7 sessions of robot-assisted shoulder-elbow mobilization (consecutive where possible, for a maximum of 5 sessions per week) in addition to standard rehabilitation. During the first and last session, the patients' residual capabilities are assessed though robotic-aided assessments as well as with clinical scales.
  Interventions: Device: Robotic treatment - NESM alpha

INTERVENTIONS:
Device: Robotic treatment - NESM alpha — The NESM-α exoskeleton can deliver passive mobilization or active-assist support that follows the patient's voluntary motion. The joints' range of motion is adjusted in each session so that the treatment is tailored to the patient's recovery. The level of assistance is tuned during the first session to be tailored on patient residual capabilities.

SUMMARY:
The study is designed as an open-label pilot study with a pre-post treatment assessment.

DETAILED DESCRIPTION:
The enrolled patients will undergo a rehabilitation program aimed at recovering upper-limb motor function. The entire cohort will receive the hospital's standard rehabilitative care, and the experimental treatment will be provided as an add-on. All participants will complete 7 sessions of robot-assisted rehabilitation (consecutive where possible, for a maximum of 5 sessions per week), with the NESM-α robotic exoskeleton. Robotic treatment consists of sessions focused on shoulder and elbow mobilization and functional movements. The range of motion is adjusted in each session so that the treatment is tailored to the patient's recovery. The level of assistance is tuned during the first session to be tailored on patient residual capabilities.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral ischemic or hemorrhagic stroke, sub-acute (<6 months) or chronic (>6 months)
* Severe spasticity (MAS ≥ 2) or mild-moderate spasticity with residual active antigravity movements (MAS < 2)
* Fugl-Meyer upper extremity score ≤ 42
* MMSE > 24
* No severe pain during passive mobilization
* Written informed consent

Exclusion Criteria:

* Unstable clinical conditions
* Inability to maintain sitting posture
* Pacemaker or other implanted electronic devices
* Passive range of motion < 10°

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2024-11-13 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | from enrollment to the end of treatment (up to 2 weeks)
  Safety of the delivered treatment is assessed monitoring the number of Adverse Events (AE). The metric is the number of events.
Feasibility of recruitment and retention | Day 7
  Evaluate the number of patients that were recruited and retained for the full study period. Evaluate the number of drop-out.

SECONDARY OUTCOMES:
Patient's functionality | Days 1 and 7
  Patient's functionality is assessed with Fugl-Meyer Assessment. It ranges from 0-66 with 0 indicating no funcionality, and 66 normal motor function.
Patient's Spasticity | Days 1 and 7
  Patient's spasticity is assessed with the Modified Ashworth Scale (MAS). It rates spasticity (muscle tone) during passive stretch.
  Range: 0, 1, 1+, 2, 3, 4. Direction: 0 = no increase in tone (best); 4 = rigid in flexion/extension (worst).
Patient's Motor Function | Days 1 and 7
  Patient's motor function is assessed with the Wolf Motor Function Test (WMFT). It assesses upper-limb motor function via 15 timed tasks plus strength measures.
  Performance Time: seconds to complete each task (often capped at 120 s if not completed). Lower = better.
Patient's Pain | Days 1 and 7
  Patient's pain is assessed with the Numeric Pain Rating Scale (NPRS). Range: 0-10 (integer or 0.5 steps). Direction: 0 = no pain (best); 10 = worst imaginable pain (worst).
Joint Angles | Days 1 and 7
  Kinematic performance of the patient using the robot is assessed with the spanned joints angles (measured in degrees)
Joint Torques | Days 1 and 7
  Kinematic performance of the patient using the robot is assessed with the joint torques (measured in Nm) exchanged with the robot

CONTACTS AND LOCATIONS:
Overall Officials: Federico Posteraro, Principal Investigator — ASL Nord Ovest Toscana
Locations (1):
- Ospedale Versilia, Lido di Camaiore, Tuscany, Italy

IPD SHARING:
Plan to Share IPD: No